CLINICAL TRIAL: NCT03474328
Title: AlcoChange: An Open Label Pilot Study of Smartphone Monitoring for Alcoholic Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Gautam Mehta, Honorary Consultant and Senior Lecturer in Hepatology, Royal Free Hospital NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16LO0290
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Alcohol-Related Disorders
MeSH Terms: conditions — Alcohol-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Device: AlcoChange

INTERVENTIONS:
Device: AlcoChange — Smartphone app and breathalyser

SUMMARY:
Alcohol contributes to over 5% of deaths worldwide, and death rates from alcohol-related liver disease (ARLD) in the UK continue to rise sharply. On-going alcohol use in ARLD leads to markedly increased mortality (Thursz et al, 2015), and maintaining abstinence is a key therapeutic goal. However, there are no effective pharmacological therapies for maintaining abstinence. Brief intervention (BI) is an effective psychological tool for reducing alcohol use, but is difficult to scale widely.

AlcoChange is a smartphone app and breathalyser (AlcoChange), which facilitates self-monitoring and delivers BIs in response to patient triggers. The aim of this open-label study is provide AlcoChange to 60 patients with ARLD, to determine compliance with the app/breathalyser and changes in self-reported alcohol consumption.

Recruitment of inpatients/outpatients with ARLD and recent alcohol use will take place at Royal Free London. The inclusion criteria are: intent to maintain abstinence, possession of compatible smartphone. The exclusion criteria are: inability to provide consent. Participants will be assessed at baseline and 3-months. The primary endpoint is self-reported alcohol use (units/week, timeline follow-back). Secondary endpoint is compliance with the app (monitored remotely).

ELIGIBILITY:
Inclusion Criteria:

* presence of ARLD
* age 18-70
* intent to maintain abstinence
* possession of compatible smartphone

Exclusion Criteria:

- inability to provide consent.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04-25 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Self-reported alcohol consumption (average/week) | 3-month study period
  Assessed by time line follow back method over study period

SECONDARY OUTCOMES:
Compliance with the app (no. of logins, duration spent on the app) | 3-month study period
  This will be assessed independently, and for associations of compliance with the app and changes in alcohol consumption (primary endpoint)